CLINICAL TRIAL: NCT03792945
Title: Comparison of the Efficacy of Corticosteroid Injection and Extracorporeal Shock Wave Therapy (ESWT) in Patients With Carpal Tunnel Syndrome; A Prospective Randomized Controlled Trial
Brief Title: Comparison of the Efficacy of Corticosteroid Injection and ESWT in Patients With CTS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ahi Evran University Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Havva Öztürk Durmaz, Research Assistant Doctor Havva ÖZTÜRK DURMAZ, Ahi Evran University Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AhiEvranUERH
Record Dates: First submitted 2018-12-07; First posted 2019-01-04 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Carpal Tunnel Syndrome; Tenosynovitis
Keywords: extracorporeal shock wave therapy; corticosteroid injection
MeSH Terms: conditions — Carpal Tunnel Syndrome; Tenosynovitis | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- extracorporeal shock wave therapy (Active Comparator): ESWT will be applied to Group 1 once a week for a total of 3 weeks. Modus ESWT device will be used. The patient's wrist will be applied at a pressure of 4 bar and 2000 Hz at a frequency of 5 Hz. Patients will be given a carpal tunnel wrist brace at night and when they do not use their hands during the day. Participants will use the carpal tunnel wrist brace 3 months.
  Interventions: Device: extracorporeal shock wave therapy
- local injection (Active Comparator): 40 mg of local Depomedrol (methylprednisolone) injection will be applied to group 2 once. Injection will be made from wrist with carpal tunnel syndrome.Patients will be given a splint at night and when they do not use their hands during the day. Participants will use the carpal tunnel wrist brace 3 months.
  Interventions: Drug: local injection
- carpal tunnel wrist brace (No Intervention): Patients will be given a carpal tunnel wrist brace at night and when they do not use their hands during the day.
  Participants will use the carpal tunnel wrist brace 3 months.

INTERVENTIONS:
Drug: local injection — In addition to the local injection, carpal tunnel brace will be given.
  Other Names: local corticosteroid injection
  Arms: local injection
Device: extracorporeal shock wave therapy — In addition to all ESWT participants, carpal tunnel brace will be given.
  Other Names: physiotheraphy
  Arms: extracorporeal shock wave therapy

SUMMARY:
In this study, the investigators aimed to demonstrate the efficacy of ESWT (extracorporeal shock wave therapy) and local corticosteroid injection in patients with carpal tunnel syndrome(CTS) compared to participants receiving only splint and exercise therapy. And the investigators wanted to show that ESWT, a noninvasive treatment modality, is as effective and reliable as local corticosteroid injection, which is the least invasive treatment. Mild and moderate CTS patients will be determined according to American Association of Electrodiagnostic Medicine (AAEM) criteria. 90 idiopathic moderate and mild CTS patients will be included in the study. The participants will be informed about their participation in a study and written informed consent will be obtained.The demographic characteristics and disease duration of the participants will be recorded.The participants will be randomly divided into 3 groups.40 mg of local methylprednisolone (depomedrol) injection will be applied to Group 1 once.

And group 1 will also be given a hand wrist rest splint to use for 3 months, especially at night, when not using the hand. ESWT will be applied to Group 2 once a week for a total of 3 weeks and hand wrist rest splints will be given for 3 months especially at night when it is not in use. Group 3 (control group) will be given a hand wrist rest splint to use for 3 months, especially at night, when not using the hand. The evaluations will be repeated before treatment, after the first week after treatment (first ESWT application) and at the 3rd month. Hand grip strength measurement will be performed using Boston carpal tunnel syndrome questionnaire, visual analog scale and dynamometer.

Electromyogram (EMG) data will be recorded before and 3 months after treatment. During the trial, the routine will not be excluded.

DETAILED DESCRIPTION:
In this study, the investigators aimed to demonstrate the efficacy of ESWT (extracorporeal shock wave therapy) and local corticosteroid injection compared to participants receiving only splint and exercise therapy. And the investigators wanted to show that ESWT, a noninvasive treatment modality, is as effective and reliable as local corticosteroid injection, which is the least invasive treatment. Mild and moderate CTS patients will be determined according to American Association of Electrodiagnostic Medicine (AAEM) criteria. Cervical radiculopathy, polyneuropathy, brachial plexopathy, systemic corticosteroid treatment, fracture and trauma history of the treated side anterior arm and wrist, inflammatory rheumatic disease, pregnant and lactating participants, participants with cardiac pacemakers, participants undergoing carpal tunnel syndrome surgery, thoracic outlet syndrome, severe atrophy, severe carpal tunnel syndrome, participants who are unwilling or unable to participate for any reason, and those who have been decided by the clinician that the participants is not in favor of the participants, systemic diseases such as renal failure, peptic ulcer, dm, hypothyroidism, coagulation disorder will be excluded.90 idiopathic moderate and mild CTS participants will be included in the study. The participants will be informed about their participation in a study and written informed consent will be obtained.The demographic characteristics and disease duration of the participants will be recorded. The participants will be randomly divided into 3 groups.40 mg of local methylprednisolone (depomedrol) injection will be applied to Group 1 once.

And group 1 will also be given a hand wrist rest splint to use for 3 months, especially at night, when not using the hand. ESWT will be applied to Group 2 once a week for a total of 3 weeks and hand wrist rest splints will be given for 3 months especially at night when it is not in use. Group 3 (control group) will be given a hand wrist rest splint to use for 3 months, especially at night, when not using the hand. The evaluations will be repeated before treatment, after the first week after treatment (first ESWT application) and at the 3rd month. Hand grip strength measurement will be performed using Boston carpal tunnel syndrome questionnaire, visual analog scale and dynamometer. Electromyogram (EMG) data will be recorded before and 3 months after treatment. During the trial, the routine will not be excluded.

ELIGIBILITY:
Inclusion Criteria:

1. Women and male patients with carpal tunnel syndrome, tendinitis, tenosynovitis diagnosed between 18-65 years of age with clinical and EMG.
2. Patients who are able to understand and correctly understand the patient information form
3. Patients consenting to participate in the study according to the informed consent form

Exclusion Criteria:

1. Cervical radiculopathy
2. Polyneuropathy
3. Brachial plexopathy
4. Systemic corticosteroid treatment
5. Fracture and trauma history of the treated side anterior arm and wrist
6. Inflammatory rheumatic disease
7. Pregnant and lactating patients
8. Patients with cardiac pacemakers
9. Patients undergoing carpal tunnel syndrome surgery
10. Thoracic outlet syndrome
11. Severe atrophy
12. Severe carpal tunnel syndrome
13. Patients who are unwilling or unable to participate for any reason, and those who have been decided by the clinician that the patient is not in favor of the patient,
14. Systemic diseases such as renal failure, peptic ulcer, dm, hypothyroidism, coagulation disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2019-04-29 (Actual); Study Completion 2019-05-29 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) - Pain | 3. months after treatment
  VAS is used to digitize some values that cannot be measured numerically.Two ends of the parameter to be evaluated are written on both ends of a 100 mm line.The participant is asked to mark the point indicating his/her status on this line.The patient marks his current state on this line.The length of the distance from where the pain is no longer to the point marked by the patient indicates the pain of the patient.The values obtained before and after treatment will be compared.The starting point of the graph is zero and the end point is 10.The distance of the point marked by the participant is measured in millimeters.And divided into 10.This value gives the participant's pain score.For example, if the point marked by the participant is 50 mm, it will get 50/10 = 5 points.Increasing the score of the participant means that the complaint is too high and the result is bad. The scale has no subscales and total score.
Visual Analog Scale (VAS) - Numbness | 3. months after treatment
  VAS is used to digitize some values that cannot be measured numerically.Two ends of the parameter to be evaluated are written on both ends of a 100 mm line. The participant is asked to mark the point indicating his / her status on this line. The patient marks his current state on this line. The length of the distance from where the numbness is no longer to the point marked by the patient indicates the numbness of the patient. The values obtained before and after treatment will be compared.The starting point of the graph is zero and the end point is 10. The distance of the point marked by the participant is measured in millimeters. And divided into 10. This value gives the participant's numbness score.For example, if the point marked by the participant is 50 mm, it will get 50/10 = 5 points.Increasing the score of the participant means that the complaint is too high and the result is bad.The scale has no subscales and total score.

SECONDARY OUTCOMES:
hand clamping force | 3. months after treatment
  Hand grip strength measurement using Jamar hydraulic hand dynamometer. Hand grip strength measurements will be performed using the elbow at 90 degrees of flexion, while the forearm and wrist is in neutral position using resistance at level 2. Measurements shall be performed three times, and the average result shall be recorded in kilograms (kg) for each hand separately.
boston scale | 3. months after treatment
  Boston symptom severity score(SSS) and improvement in functional status score(FSS). There are 11 questions at SSS. Responses vary from 'none(1 point)' to 'very severe(5 points)'. There are 8 questions in FSS. Responses vary from 'very easy (1 point)' to 'very difficult (5 points) according to difficulty level. In both scales, the degree of symptom severity and dysfunction increases as the total score increases.The score of the patient is divided by the total score (total score is 11x5 = 55 for the SSS and the total score is 8x5 = 40 for FSS) and 0 to 1 for each patient. As this ratio reaches 1, the degree of symptom severity and dysfunction of the patient increases. For example; Considering that the total score obtained from all the questions in the SPS is 22, the ratio of 22/55 = 0. 4 is obtained.These scales will be applied after treatment and the rates obtained before and after treatment will be compared.
Median nerve sensory distal latency(electrophysiological examination,physiological parameter) | 3. months after treatment
  Evaluation of median nerve sensory distal latency: Active and reference electrodes in the form of superficial electrodes will be placed in the metacarpophalangial and distal interphalangial joints of the 2nd finger. On EMG examination, sensory distal latency was greater than 3.6 ms and CTS was accepted.
Median nerve sensory transmission rate( electrophysiological examination, physiological parameter) | 3. months after treatment
  Evaluation of median nerve sensory transmission rate: Active and reference electrodes in the form of superficial electrodes will be placed in the metacarpophalangial and distal interphalangial joints of the 2nd finger. Emotional nerve conduction velocity lower than 50 m/s in EMG examination will be accepted as CTS.
Median nerve motor distal latency( electrophysiological examination, physiological parameter) | 3. months after treatment
  Evaluation of median nerve motor distal latency : The patient will be stretched in the supine position with the arm extended, the palm facing up.The active recording electrode will be connected to the middle point of the abductor pollicis brevis (APB), the reference electrode to the thumb, the ground electrode to the flexor face of the forearm.The first warning will be given by the ulnar of the brachial artery pulse from the proximal 5 cm proximal part of the active electrode to the wrist. In the EMG examination, if the motor distal latency is over 4.2 ms, CTS will be accepted.
Median nerve motor transmission rate ( electrophysiological examination, physiological parameter) | 3. months after treatment
  Evaluation of median nerve motor transmission rate: The patient will be stretched in the supine position with the arm extended, the palm facing up.The active recording electrode will be connected to the middle point of the abductor pollicis brevis (APB), the reference electrode to the thumb, the ground electrode to the flexor face of the forearm.The first warning will be given by the ulnar of the brachial artery pulse from the proximal 5 cm proximal part of the active electrode to the wrist.
Median sensory nerve action potential amplitude | 3. months after treatment
  Evaluation of Median sensory nerve action potential amplitude: Active and reference electrodes in the form of superficial electrodes will be placed in the metacarpophalangial and distal interphalangial joints of the 2nd finger. In the emg examination, the median sensory nerve action potential amplitude below 10 microvolts will be accepted as CTS.
Compound muscle action potential amplitude | 3. months after treatment
  Evaluation of compound muscle action potential amplitude: The patient will be stretched in the supine position with the arm extended, the palm facing up.The active recording electrode will be connected to the middle point of the abductor pollicis brevis (APB), the reference electrode to the thumb, the ground electrode to the flexor face of the forearm.The first warning will be given by the ulnar of the brachial artery pulse from the proximal 5 cm proximal part of the active electrode to the wrist. The median CBAP amplitude below 5 millivolt in the recording of APB muscle in the emg examination will be accepted as CTS.

CONTACTS AND LOCATIONS:
Overall Officials: Havva ÖZTÜRK DURMAZ, Principal Investigator — Ahi Evran University Education and Research Hospital
Locations (1):
- Ahi Evran University Education and Research Hospital, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozturk Durmaz H, Tuncay F, Durmaz H, Erdem HR. Comparison of Radial Extracorporeal Shock Wave Therapy and Local Corticosteroid Injection Effectiveness in Patients With Carpal Tunnel Syndrome: A Randomized Controlled Study. Am J Phys Med Rehabil. 2022 Jul 1;101(7):685-692. doi: 10.1097/PHM.0000000000001891. Epub 2021 Oct 4. PMID 35706121